CLINICAL TRIAL: NCT06990100
Title: Clinical Performance and Safety of ENDOPACK® DT4-EBMCA in ACL Reconstruction 24 Months Post-surgery : Post-market Clinical Follow-up Study
Acronym: DT4-EBMCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SACIMEX (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A01222-45
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: ACL Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACL rupture group (Active Comparator): Patients having a surgery with DT4-EBMCA medical device
  Interventions: Device: ACL surgery

INTERVENTIONS:
Device: ACL surgery — ligamentoplasty surgery - ACL reconstruction surgery

SUMMARY:
Anterior cruciate ligament (ACL) injuries are among the most common sports-related knee traumas. The DT4-EBMCA device, based on a quadrupled semitendinosus autograft technique, aims to provide effective and minimally invasive ligament reconstruction. This study evaluates its long-term performance and safety in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with DT4-EBMCA in Médipôle Garonne for a total or partial rupture of the anterior cruciate ligaments
* Patient having answer to IKDC and KOOS pre-operative
* Patient having received information and signed informed consent

Exclusion Criteria:

* Patients who refuse to participate
* Patients unable to understand questionnaires
* Patients who, at the time of surgery, present the contraindications and Factors likely to jeopardize the success of the implant contained in the IFU :
* Acute or chronic, local or systemic infections;
* Severe muscular, neurological or vascular impairments affecting the extremity concerned;
* Bone destruction or poor bone quality that may affect device stability;
* Any concomitant condition that may affect device function;
* Patients with sensitivity to device material that may cause allergic reactions.
* Severe osteoporosis;
* Significant deformity, congenital dislocation;
* Local bone tumours;
* Systemic or metabolic disorders;
* Infectious diseases;
* Substance abuse and/or tendencies to abuse drugs or medication;
* Obesity;
* Unsupervised intense physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
evaluate the performance of the DT4- EBMCA | 2 years post-surgery
  International Knee Documentation Committee (IKDC) from the preoperative visit to the postoperative 2 years follow-up Knee injury and Osteoarthritis Outcome Score (KOOS) from the preoperative visit to the postoperative 2 years follow-up

SECONDARY OUTCOMES:
safety of of the DT4-EBMCA | 2 years post-surgery
  Mean rate of complications from the preoperative visit to the postoperative 2 years follow-up Re-rupture ≤ 2,5%

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique MEDIPOLE GARONNE, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided